CLINICAL TRIAL: NCT06958861
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Inhaled H057 in the Treatment of Acute Exacerbations of Bronchiectasis
Brief Title: A Clinical Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Inhaled H057 in the Treatment of Acute Exacerbations of Bronchiectasis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Huilun Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PH-H057-II-03
Record Dates: First submitted 2025-04-16; First posted 2025-05-06 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Acute Exacerbations of Bronchiectasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose H057+standard-of-care (Experimental): Subjects are administered low-dose inhaled H057, combined with standard-of-care treatment, which included anti-infective therapy, expectorant therapy, hemostasis, oxygen therapy, and other supportive measures.
  Interventions: Drug: Low-dose H057+standard-of-care
- High dose H057+standard-of-care (Experimental): Subjects are administered high-dose inhaled H057, combined with standard-of-care treatment, which included anti-infective therapy, expectorant therapy, hemostasis, oxygen therapy, and other supportive measures.
  Interventions: Drug: High-dose H057+standard-of-care
- H057 placebo+standard-of-care (Placebo Comparator): Subjects are administered inhaled H057 placebo, combined with standard-of-care treatment, which included anti-infective therapy, expectorant therapy, hemostasis, oxygen therapy, and other supportive measures.
  Interventions: Drug: H057 placebo+standard-of-care

INTERVENTIONS:
Drug: Low-dose H057+standard-of-care — Subjects are administered low-dose inhaled H057, combined with standard-of-care treatment, which included anti-infective therapy, expectorant therapy, hemostasis, oxygen therapy, and other supportive measures.
  Arms: Low dose H057+standard-of-care
Drug: High-dose H057+standard-of-care — Subjects are administered high-dose inhaled H057, combined with standard-of-care treatment, which included anti-infective therapy, expectorant therapy, hemostasis, oxygen therapy, and other supportive measures.
  Arms: High dose H057+standard-of-care
Drug: H057 placebo+standard-of-care — Subjects are administered inhaled H057 placebo, combined with standard-of-care treatment, which included anti-infective therapy, expectorant therapy, hemostasis, oxygen therapy, and other supportive measures.
  Arms: H057 placebo+standard-of-care

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled trial to evaluate the efficacy, safety, pharmacokinetics, and pharmacodynamics of inhaled H057 in the treatment of acute exacerbations of bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be eligible for enrollment in this study:

1. Age ≥18 years, regardless of gender;
2. Patients who are determined by the investigator to be in an acute exacerbation phase of bronchiectasis prior to enrollment: at least three out of the following six symptoms-cough, changes in sputum volume, purulent sputum, dyspnea or reduced exercise tolerance, fatigue or malaise, hemoptysis-have worsened for more than 48 hours, and the clinician deems that intervention is necessary;
3. Able to tolerate nebulized inhalation treatment;
4. After instruction, able to correctly use the nebulizer for treatment and accurately complete questionnaires;
5. Subjects must fully understand the purpose, nature, methods, and potential adverse events of the trial, voluntarily agree to participate, and sign the informed consent form, or have a legally authorized representative provide informed consent on their behalf.

Exclusion Criteria:

If a subject meets any of the following criteria, they are not eligible to participate in this study:

1. Patients with bronchiectasis caused by cystic fibrosis, as determined by the investigator;
2. Patients who have experienced an acute exacerbation of bronchiectasis for more than 7 days;
3. Patients with an acute exacerbation of bronchiectasis who have received intravenous antibiotic treatment for more than 72 hours prior to enrollment;
4. Patients with mild bronchiectasis caused by asthma;
5. Patients with comorbid allergic bronchopulmonary aspergillosis, active tuberculosis, or active non-tuberculous mycobacterial infection requiring standardized treatment;
6. Patients with moderate or massive hemoptysis during an acute exacerbation of bronchiectasis (moderate hemoptysis: 100-500 mL within 24 hours; massive hemoptysis: >500 mL within 24 hours or a single episode of 100-500 mL);
7. Patients with significant liver or kidney dysfunction (ALT, AST >2 times the upper limit of normal [ULN]; Cr >1.5 times ULN);
8. Patients with a history of malignancy or who have achieved clinical remission for less than 5 years;
9. Patients with any other unstable clinical conditions deemed significant by the investigator, including but not limited to cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, psychiatric, or major physiological dysfunction, and: a) Whose condition may affect the patient's safety during the study; b) That may impact the study results and their interpretation; c) That may hinder the patient's ability to complete the entire study;
10. Patients who are positive for hepatitis B surface antigen (HBsAg) with HBV-DNA >1000 copies/mL or 200 IU/mL, or positive for hepatitis C virus antibody (HCV-Ab), human immunodeficiency virus antibody (HIV-Ab), or anti-Treponema pallidum antibody;
11. Patients who are allergic to the active ingredients or excipients of the investigational product or who have a history of hypersensitivity or an allergic constitution;
12. Patients who have participated in other drug or medical device trials within the past 3 months or are currently participating in another clinical trial;
13. Pregnant women, lactating women, and women of childbearing potential;
14. Subjects whom the investigator considers unsuitable for participation in this study for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Quality-of-Life Bronchiectasis Respiratory Symptom Score | baseline to day 15
  To evaluate change in Quality-of-Life Bronchiectasis Respiratory Symptom Score (QoL-B-RSS) from baseline.
  QoL-B-RSS, a self-administered, patient-reported outcome measure assessing symptoms, functioning and health-related quality of life for patients with non-cystic fibrosis (CF) bronchiectasis, contains 37 items on 8 scales (Respiratory Symptoms, Physical, Role, Emotional and Social Functioning, Vitality, Health Perceptions and Treatment Burden). It scores ranging from 0 to 100, where lower scores indicated more severe symptoms.

SECONDARY OUTCOMES:
Quality-of-Life Bronchiectasis Respiratory Symptom Score | baseline to day 29 or day 1 post-treatment
  To evaluate change in Quality-of-Life Bronchiectasis Respiratory Symptom Score (QoL-B-RSS) from baseline.
  QoL-B-RSS, a self-administered, patient-reported outcome measure assessing symptoms, functioning and health-related quality of life for patients with non-cystic fibrosis (CF) bronchiectasis, contains 37 items on 8 scales (Respiratory Symptoms, Physical, Role, Emotional and Social Functioning, Vitality, Health Perceptions and Treatment Burden). It scores ranging from 0 to 100, where lower scores indicated more severe symptoms.
treatment efficacy rate | baseline to day 15
  Response to treatment is defined as the significant improvement or near resolution of acute exacerbation symptoms.
  Treatment failure is defined as the absence of significant improvement or progressive worsening of acute exacerbation symptoms, such as requiring hospitalization or the need for additional antibiotic therapy.
clinical pulmonary infection score | baseline to day 15
  To evaluate change in clinical pulmonary infection score (CPIS) from baseline. The CPIS is calculated on the basis of points assigned for various signs and symptoms of pneumonia (eg, fever and extent of oxygenation impairment). It scores ranging from 0 to 12, where higher scores mean a worse outcome. Some studies suggest that a CPIS >6 may correlate with ventilator-associated pneumonia (VAP).
bronchiectasis exacerbation and symptom tool | baseline to day 29 or day 1 post-treatment
  To evaluate change in bronchiectasis exacerbation and symptom tool (BEST) from baseline.
  The BEST diary is to detect bronchiectasis exacerbations. It scores ranging from 0 to 26, where higher scores indicate more severe symptoms.The BEST symptom diary is responsive at onset and recovery from exacerbation and may be useful to capture and characterise exacerbations.
Borg Scale | baseline to day 29 or day 1 post-treatment
  To evaluate change in Borg Scale from baseline. Borg Scale is one of commonly used measures to assess dyspnea in chronic lung disease.The scale was modified to form a 10-point scale including written indicators of severity. The scale has been used to quantify various "perceived symptoms" such as breathlessness and muscle fatigue during exercise. The higher Borg Scale means more severe breathlessness and muscle fatigue
sputum purulence score | baseline to day 29 or day 1 post-treatment
  To evaluate change in sputum purulence score from baseline. It scores ranging from 0 to 8, where a higher score indicates greater severity of the condition.
24-hour sputum volume | baseline to day 29 or day 1 post-treatment
  To evaluate change in 24-hour sputum volume from baseline
FEV1%pred | baseline to day 29 or day 1 post-treatment
  To evaluate change in FEV1%pred from baseline
the frequency of acute exacerbations in bronchiectasis | day 1 to day 180
safety of inhaled H057 in acute exacerbations of bronchiectasis | day 1 to day 180
  the incidence and severity of adverse events (AEs) and serious adverse events (SAEs), as well as changes in vital signs and laboratory test results, etc.
pharmacokinetic characteristics--Cmax | day 1 to day 28
pharmacokinetic characteristics--Tmax | day 1 to day 28
pharmacokinetic characteristics--t1/2 | day 1 to day 28
pharmacokinetic characteristics--AUC0-t | day 1 to day 28
pharmacokinetic characteristics--Rac | day 1 to day 28
pharmacodynamic characteristic | day 1 to day 28
  To evaluate change in neutrophil elastase levels from baseline

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - Fuyang Hospital Of Anhui Medical University, Fuyang, Anhui
  - Hefei First People's Hospital, Hefei, Anhui
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Affiliated hospital of Youjiang Medical University For Nationalities, Baise City, Guangxi
  - Hebei General Hospital, Shijiazhuang, Hebei
  - Nanyang Second General Hospital, Nanyang, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - The second Xiangya Hospital of Central South University, Changsha, Hunan
  - Changzhou First People's Hospital, Changzhou, Jiangsu
  - Jiujiang No.1 People's Hospital, Jiujiang, Jiangxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Deyang People's Hospital, Deyang, Sichuan
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Jinhua Municipal Central Hospital, Jinhua, Zhejiang
  - Ningbo No.2 Hospital, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang